CLINICAL TRIAL: NCT01532570
Title: To Evaluate the Efficacy, Safety, and Pharmacokinetics of TA-650 in Patients With Behcet's Disease ( BD ) With Special Lesions After the Administration of TA-650
Brief Title: Clinical Study of TA-650 in Patients With Behcet's Disease (BD) With Special Lesions
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TA-650-23
Record Dates: First submitted 2012-02-06; First posted 2012-02-14 (Estimated); Results first posted 2016-12-16 (Estimated); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Behcet's Disease; Behcet Syndrome; Neuro-Behcet's Disease
Keywords: Behcet's disease; intestinal Behcet's disease; neuro-Behcet's disease; vascular Behcet's disease
MeSH Terms: conditions — Behcet Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TA-650 (Experimental)
  Interventions: Drug: TA-650

INTERVENTIONS:
Drug: TA-650 — TA-650 will be intravenously infused at a dosage of 5 mg/kg slowly over a period of more than 2 hours at the first administration (weeks 0), 2, and 6, and then every 8 weeks up to week 46. If the criteria for a dosage escalation are met at the evaluation after week 30, TA-650 will be administered at a dosage of 10 mg/kg after week 30.

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety, and pharmacokinetics of TA-650 in patients with Behcet's disease ( BD ) with special lesions after the administration of TA-650 at a dosage of 5 mg/kg in weeks 0, 2, and 6, then every 8 weeks after week 14 up to week 46.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were diagnosed with the complete or incomplete type of Behcet's disease according to "The criteria for a diagnosis of Behcet's disease, Ministry of Health, Labour and Welfare in Japan (partially revised in 2010)"
* Patients who have special lesions despite having received conventional treatments for special lesions, or patients who cannot receive conventional treatments due to intolerability.
* Patients who have clinical symptoms associated with each special lesions.

Exclusion Criteria:

* Patients with intestinal, neuro-, vascular Behcet's disease in whom a differential diagnosis of each Behcet's disease from other conditions．
* Patients who have received treatment with infliximab within 1 year before enrollment for another purpose than treating special lesions; or patients whose previous treatment with infliximab was discontinued due to adverse events.
* Patients who had participated in another clinical study and had received a study drug within 12 weeks before giving acquirement.

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2012-01; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yoshiaki Ishigatsubo, MD, Ph.D, Study Director — Yokohama City University Graduate School of Medicine; Toshifumi Hibi, MD, Study Director — Kitasato University Kitasato Institute Hospital; Shunsei Hirohata, MD, Study Director — Kitasato University School of Medicine; Kazuoki Kondo, MD, Study Director — Mitsubihsi Tanabe Pharma Corporation
Locations (6):
- Japan (6):
  - Investigational site, Chūbu
  - Investigational site, Hokkaido
  - Investigational site, Kanto
  - Investigational site, Kinki
  - Investigational site, Kyusyu
  - Investigational site, Tōhoku

REFERENCES:
- [Result] Hibi T, Hirohata S, Kikuchi H, Tateishi U, Sato N, Ozaki K, Kondo K, Ishigatsubo Y. Infliximab therapy for intestinal, neurological, and vascular involvement in Behcet disease: Efficacy, safety, and pharmacokinetics in a multicenter, prospective, open-label, single-arm phase 3 study. Medicine (Baltimore). 2016 Jun;95(24):e3863. doi: 10.1097/MD.0000000000003863. PMID 27310969

RESULTS

PARTICIPANT FLOW:
Groups:
- Intestinal BD; Acute Neuro-BD; Chronic Progressive Neuro-BD; Vascular BD: A-650, 5 mg/kg, iv infusion over a period of more than 2 hours. If the criteria for a dosage escalation are met at the evaluation after week 30, TA-650 will be administered at a dosage of 10 mg/kg after week 30.
Period: Overall Study
Arm/Group | Intestinal BD | Acute Neuro-BD | Chronic Progressive Neuro-BD | Vascular BD
Started | 11 | 2 | 1 | 4
Completed | 10 | 1 | 1 | 4
Not Completed | 1 | 1 | 0 | 0
Not completed — Lack of Efficacy | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intestinal BD | Acute Neuro-BD | Chronic Progressive Neuro-BD | Vascular BD | Total
Number analyzed (Participants) | 11 | 2 | 1 | 4 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.0 (13.4) | 34.0 (5.7) | 47.0 (NA) — There is no data because the Overall Number of Baseline Participant is 1. | 44.0 (2.9) | 37.6 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 1 | 0 | 1 | 8
  Male | 5 | 1 | 1 | 3 | 10

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Complete Response at Week 30
Description: We defined the patient who met the following criteria as the complete responders.
  The criteria of complete responders are that clinical symptoms associated with each BD have disappeared and morphological characteristics (ex. ulcers area, Computed tomography (CT) or Positron emission tomography/Computed tomography (PET/CT) findings etc) at the lesion site and inflammatory markers (ex. cerebrospinal fluid and serum inflammatory markers) are improved compared to Week 0.
Time Frame: Week 30
Measure: Number; unit: percentage of Complete Responders
Arm/Group | Intestinal BD | Acute Neuro-BD | Chronic Progressive Neuro-BD | Vascular BD
Number analyzed (Participants) | 11 | 2 | 1 | 4
percentage of Complete Responders | 54.5 | 0 | 100 | 100

2. Secondary Outcome: Percentage of Participants With Complete Response at Week 14 and 54
Description: We defined the patient who met the following criteria as the complete responders.
  The criteria of complete responders are that clinical symptoms associated with each BD have disappeared and morphological characteristics (ex. ulcers area, CT or PET/CT findings etc) at the lesion site and inflammatory markers (ex. cerebrospinal fluid and serum inflammatory markers) are improved compared to Week 0.
Time Frame: Week 14, Week 54
Measure: Number; unit: percentage of Complete Responders
Arm/Group | Intestinal BD | Acute Neuro-BD | Chronic Progressive Neuro-BD | Vascular BD
Number analyzed (Participants) | 11 | 2 | 1 | 4
percentage of Complete Responders
  Week 14 (n=11, 2, 1, 4) | 54.5 | 0 | 100 | 100
  Week 54 (n=10, 1, 1, 4) | 60 | 0 | 100 | 100

3. Secondary Outcome: Patient General Visual Analogue Scale (VAS) for the Clinical Symptoms Associated With Each BD
Description: The VAS evaluation measured using the "General VAS evaluation From" and the range is from 0 to 100 mm. The best condition per one week before evaluation visit for the clinical symptoms associated with each BD is defined as "0" and the worst condition is defined as "100".
  The time of final evaluation : Final time point for the 5 mg/kg patients, final time point during administration of 5 mg/kg for the 10 mg/kg patients, final time point during administration of 5 mg/kg for patients who discontinued the study.
Time Frame: Week 0, 2, 6, 10, then every 4 weeks after Week 14 to Week 54
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Neuro-BD (Acute+Chronic Progressive): Acute; A-650, 5 mg/kg, iv infusion over a period of more than 2 hours. If the criteria for a dosage escalation are met at the evaluation after week 30, TA-650 will be administered at a dosage of 10 mg/kg after week 30.
  Chronic Progressive; A-650, 5 mg/kg, iv infusion over a period of more than 2 hours. If the criteria for a dosage escalation are met at the evaluation after week 30, TA-650 will be administered at a dosage of 10 mg/kg after week 30.
Arm/Group | Intestinal BD | Neuro-BD (Acute+Chronic Progressive) | Vascular BD
Number analyzed (Participants) | 11 | 3 | 4
units on a scale
  Week 0 (n=11, 3, 4) | 55.5 (22.9) | 41.3 (11.0) | 40.5 (34.4)
  Week 2 (n=11, 3, 4) | 42.7 (30.9) | 33.0 (23.1) | 11.8 (7.8)
  Week 6 (n=11, 3, 4) | 26.4 (20.3) | 15.0 (17.1) | 14.3 (8.1)
  Week 10 (n=11, 3, 4) | 23.6 (19.8) | 23.0 (20.4) | 17.8 (14.0)
  Week 14 (n=11, 3, 4) | 32.4 (24.0) | 28.3 (30.0) | 13.5 (9.8)
  Week 18 (n=11, 3, 4) | 23.9 (20.8) | 31.7 (22.4) | 15.3 (8.9)
  Week 22 (n=11, 3, 4) | 31.8 (26.0) | 35.3 (31.5) | 17.8 (6.4)
  Week 26 (n=11, 2, 4) | 28.9 (20.7) | 18.5 (23.3) | 17.5 (9.8)
  Week 30 (n=11, 2, 4) | 31.1 (29.2) | 15.0 (21.2) | 11.8 (7.5)
  Week 34 (n=11, 2, 4) | 21.2 (21.6) | 12.5 (17.7) | 18.8 (9.2)
  Week 38 (n=11, 2, 4) | 25.4 (30.8) | 11.5 (16.3) | 10.3 (8.3)
  Week 42 (n=10, 2, 4) | 20.9 (20.4) | 13.0 (18.4) | 13.5 (9.3)
  Week 46 (n=10, 2, 4) | 22.3 (27.5) | 11.5 (16.3) | 10.5 (6.6)
  Week 50 (n=10, 2, 4) | 17.5 (25.1) | 11.5 (16.3) | 22.8 (25.4)
  Week 54 (n=10, 2, 4) | 21.0 (26.6) | 8.5 (12.0) | 11.3 (7.9)
  Final (n=11, 3, 4) | 26.9 (29.6) | 7.7 (8.6) | 11.3 (7.9)

4. Secondary Outcome: Imaging Findings:Endoscopic Examination for Intestinal BD
Description: The investigator assessed the length of the major axis of the principal intestinal ulcer at day of evaluation and scored in accordance with the following categories, "Healed/scarred, Reduced to =< 25%, Reduced to > 25% to =< 50% or Reduced to > 50%/no change/increased" in the principal intestinal ulcer compared to size at Week 0.
Time Frame: Week 14, Week 30, Week 54
Measure: Number; unit: participants
Arm/Group | Intestinal BD
Number analyzed (Participants) | 11
participants
  The ulcer was cured or scarred: Week 14 (n=11) | 9
  Reduced to = < 1/4: Week 14 (n=11) | 0
  Reduced to > 1/4 to = < 1/2: Week 14 (n=11) | 0
  Reduced to > 1/2 or increase: Week 14 (n=11) | 2
  The ulcer was cured or scarred: Week 30 (n=11) | 9
  Reduced to = < 1/4: Week 30 (n=11) | 0
  Reduced to > 1/4 to = < 1/2: Week 30 (n=11) | 0
  Reduced to > 1/2 or increase: Week 30 (n=11) | 2
  The ulcer was cured or scarred: Week 54 (n=9) | 8
  Reduced to = < 1/4: Week 54 (n=9) | 0
  Reduced to > 1/4 to = < 1/2: Week 54 (n=9) | 0
  Reduced to > 1/2 or increase: Week 54 (n=9) | 1
  The ulcer was cured or scarred: Final (n=11) | 9
  Reduced to = < 1/4: Final (n=11) | 0
  Reduced to > 1/4 to = < 1/2: Final (n=11) | 0
  Reduced to > 1/2 or increase: Final (n=11) | 2

5. Secondary Outcome: Imaging Findings: Brain Magnetic Resonance Imaging (MRI) for Acute Neuro-BD
Description: Changes in brain MRI findings were scored at day of evaluation, in accordance with the following categories, "No high-intensity areas, Reduction or No changes/increase" in the size of high-intensity areas compared to Week 0.
Time Frame: Week 14, Week 30, Week 54
Measure: Number; unit: participants
Arm/Group | Acute Neuro-BD
Number analyzed (Participants) | 2
participants
  Reduced high intensity areas, Week 14 (n=2) | 2
  Reduced high intensity areas, Week 30 (n=1) | 1
  Reduced high intensity areas, Week 54 (n=1) | 1

6. Secondary Outcome: Imaging Findings: Brainstem MRI for Chronic Neuro-BD
Description: Changes in brainstem MRI findings were scored at day of evaluation, in accordance with the following categories, "Unchanged or Reduced" in the brainstem area compared to Week 0.
Time Frame: Week 14, Week 30, Week 54
Measure: Number; unit: participants
Arm/Group | Chronic Progressive Neuro-BD
Number analyzed (Participants) | 1
participants
  Unchanged brain stem area, Week 14 | 1
  Unchanged brain stem area, Week 30 | 1
  Unchanged brain stem area, Week 54 | 1

7. Secondary Outcome: Imaging Findings: CT, PET/CT for Vascular-BD
Description: Changes in CT or PET/CT findings were scored at day of evaluation, in accordance with the following categories, "Improves, Unchanged or Worsened" by comparison with those at Week 0.
Time Frame: Week 14, Week 30, Week 54
Measure: Number; unit: participants
Groups:
- Vascular-BD: A-650, 5 mg/kg, iv infusion over a period of more than 2 hours. If the criteria for a dosage escalation are met at the evaluation after week 30, TA-650 will be administered at a dosage of 10 mg/kg after week 30.
Arm/Group | Vascular-BD
Number analyzed (Participants) | 4
participants
  Improved, Week 14 | 3
  Unchanged, Week 14 | 1
  Woesened, Week 14 | 0
  Improved, Week 30 | 3
  Unchanged, Week 30 | 1
  Worsened, Week 30 | 0
  Improved, Week 54 | 3
  Unchanged, Week 54 | 1
  Worsened, Week 54 | 0

8. Secondary Outcome: Concentration of Inflammatory Biomarker (C-reactive Protein (CRP)) of Intestinal BD
Description: The time of final evaluation : Final time point for the 5 mg/kg patients, final time point during administration of 5 mg/kg for the 10 mg/kg patients, final time point during administration of 5 mg/kg for patients who discontinued the study.
Time Frame: Week 0, 2, 6, 10, then every 4 weeks after Week 14 to Week 54
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Intestinal BD
Number analyzed (Participants) | 11
mg/dL
  Week 0 (n=11) | 0.20 [0.00 to 1.00]
  Week 2 (n=11) | 0.00 [0.00 to 0.00]
  Week 6 (n=11) | 0.10 [0.00 to 0.10]
  Week 10 (n=11) | 0.10 [0.00 to 0.30]
  Week 14 (n=10) | 0.15 [0.00 to 0.80]
  Week 18 (n=11) | 0.10 [0.00 to 0.10]
  Week 22 (n=11) | 0.10 [0.00 to 0.50]
  Week 26 (n=11) | 0.00 [0.00 to 0.10]
  Week 30 (n=11) | 0.10 [0.00 to 2.20]
  Week 34 (n=11) | 0.00 [0.00 to 0.30]
  Week 38 (n=11) | 0.10 [0.00 to 0.60]
  Week 42 (n=10) | 0.00 [0.00 to 0.20]
  Week 46 (n=10) | 0.00 [0.00 to 0.10]
  Week 50 (n=10) | 0.05 [0.00 to 0.10]
  Week 54 (n=10) | 0.10 [0.00 to 0.20]
  Final (n=11) | 0.10 [0.00 to 0.20]

9. Secondary Outcome: Concentration of Inflammatory Biomarker (CRP) of Vascular BD
Description: as for outcome 8
Time Frame: Week 0, 2, 6, 10, then every 4 weeks after Week 14 to Week 54
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Vascular-BD
Number analyzed (Participants) | 4
mg/dL
  Week 0 | 0.90 [0.55 to 2.65]
  Week 2 | 0.25 [0.10 to 0.35]
  Week 6 | 0.20 [0.05 to 0.30]
  Week 10 | 0.10 [0.05 to 0.10]
  Week 14 | 0.15 [0.10 to 0.30]
  Week 18 | 0.15 [0.10 to 0.25]
  Week 22 | 0.10 [0.10 to 0.10]
  Week 26 | 0.10 [0.10 to 0.15]
  Week 30 | 0.10 [0.05 to 0.15]
  Week 34 | 0.10 [0.05 to 0.25]
  Week 38 | 0.15 [0.10 to 0.85]
  Week 42 | 0.10 [0.10 to 0.15]
  Week 46 | 0.15 [0.10 to 0.20]
  Week 50 | 0.05 [0.00 to 1.05]
  Week 54 | 0.15 [0.05 to 0.20]
  Final | 0.15 [0.05 to 0.20]

10. Secondary Outcome: Level of Inflammatory Biomarker (Erythrocyte Sedimentation Rate) of Vascular BD
Description: as for outcome 8
Time Frame: Week 0, 2, 6, 10, then every 4 weeks after Week 14 to Week 54
Measure: Median (Inter-Quartile Range); unit: mm/hr
Arm/Group | Vascular-BD
Number analyzed (Participants) | 4
mm/hr
  Week 0 | 31.0 [21.5 to 35.5]
  Week 2 | 11.0 [7.0 to 14.5]
  Week 6 | 8.0 [3.0 to 12.5]
  Week 10 | 7.0 [3.0 to 11.0]
  Week 14 | 8.5 [3.5 to 13.0]
  Week 18 | 6.5 [3.0 to 11.0]
  Week 22 | 5.5 [3.0 to 11.0]
  Week 26 | 7.5 [2.5 to 11.0]
  Week 30 | 4.5 [4.0 to 9.5]
  Week 34 | 6.5 [2.5 to 13.0]
  Week 38 | 9.0 [5.0 to 11.0]
  Week 42 | 9.5 [5.5 to 11.0]
  Week 46 | 8.5 [4.5 to 10.5]
  Week 50 | 8.0 [5.0 to 10.5]
  Week 54 | 6.5 [3.0 to 9.0]
  Final | 6.5 [3.0 to 9.0]

11. Secondary Outcome: Cell Counts in Cerebrospinal Fluid (CSF) for Acute Neuro-BD
Description: as for outcome 8
Time Frame: Week 0, Week 14, Week 30, Week 54
Measure: Number; unit: cells/mL
Arm/Group | Acute Neuro BD (Patient 1) | Acute Neuro-BD (Patient 2)
Number analyzed (Participants) | 1 | 1
cells/mL
  Week 0 | 37 | 3
  Week 14 | 4 | 2
  Week 30 | 1 | NA — There is no data because of discontinuation
  Week 54 | NA — The value is Limit of Quantification (LOQ)) (i.e. =<1) | NA — There is no data because of discontinuation
  At discontinuation | NA — There is no data because of completion | 2

12. Secondary Outcome: Interleukin-6 (IL-6) Concentration in CSF for Neuro-BD
Time Frame: Week 0, Week 14, Week 30, Week 54
Measure: Number; unit: pg/mL
Arm/Group | Acute Neuro BD (Patient No.1) | Acute Neuro-BD (Patient No.2) | Chronic Progressive Neuro-BD
Number analyzed (Participants) | 1 | 1 | 1
pg/mL
  Week 0 | 145 | 2.5 | 64.5
  Week 14 | 2.2 | 23 | 35.1
  Week 30 | 1.4 | NA — There is no data because of discontinuation | 5.4
  Week 54 | 1.5 | NA — There is no data because of discontinuation | 32.1
  At discontinuation | NA — There is no data because of completion | 6.5 | NA — There is no data because of completion

13. Secondary Outcome: The Number of Improved Intestinal BD Patients From Baseline
Description: The investigator assessed clinical symptoms associated with intestinal BD in one week before the day of evaluation as " No symptom, Very slightly poor, Slightly poor, Poor or Extremely poor".
  We calculated improved patients in comparison with those for Week 0.
Time Frame: Week 0, 2, 6, 10, then every 4 weeks after Week 14 to Week 54
Measure: Number; unit: participants
Arm/Group | Intestinal BD
Number analyzed (Participants) | 11
participants
  Week 2 (n=11) | 7
  Week 6 (n=11) | 9
  Week 10 (n=11) | 9
  Week 14 (n=11) | 8
  Week 18 (n=11) | 11
  Week 22 (n=11) | 10
  Week 26 (n=11) | 10
  Week 30 (n=11) | 10
  Week 34 (n=11) | 10
  Week 38 (n=11) | 9
  Week 42 (n=10) | 8
  Week 46 (n=10) | 8
  Week 50 (n=10) | 8
  Week 54 (n=10) | 8
  Final (n=11) | 9

14. Secondary Outcome: Change From Baseline in Clinical Symptoms Associated With Neuro-BD Patients
Description: The investigator assessed the clinical symptoms associated with neuro-BD at each time point of the evaluation in compared to Week 0, in accordance with the categories as "No symptom, Improved, Unchanged or Worsened".
Time Frame: Week 2, 6, 10, then every 4 weeks after Week 14 to Week 54
Measure: Number; unit: participants
Arm/Group | Acute Neuro BD (Patient No.1) | Acute Neuro-BD (Patient No.2) | Chronic Progressive Neuro-BD
Number analyzed (Participants) | 1 | 1 | 1
participants
  No symptom, Week 2 | 1 | 1 | 0
  Improved, Week 2 | 0 | 0 | 0
  Unchanged, Week 2 | 0 | 0 | 1
  Worsened, Week 2 | 0 | 0 | 0
  No symptom, Week 6 | 1 | 1 | 1
  Improved, Week 6 | 0 | 0 | 0
  Unchanged, Week 6 | 0 | 0 | 0
  Worsened, Week 6 | 0 | 0 | 0
  No symptom, Week 10 | 1 | 0 | 0
  Improved, Week 10 | 0 | 1 | 1
  Unchanged, Week 10 | 0 | 0 | 0
  Worsened, Week 10 | 0 | 0 | 0
  No symptom, Week 14 | 1 | 0 | 1
  Improved, Week 14 | 0 | 1 | 0
  Unchanged, Week 14 | 0 | 0 | 0
  Worsened, Week 14 | 0 | 0 | 0
  No symptom, Week 18 | 1 | 0 | 1
  Improved, Week 18 | 0 | 1 | 0
  Unchanged, Week 18 | 0 | 0 | 0
  Worsened, Week 18 | 0 | 0 | 0
  No symptom, Week 22 | 0 | 0 | 1
  Improved, Week 22 | 1 | 0 | 0
  Unchanged, Week 22 | 0 | 1 | 0
  Worsened, Week 22 | 0 | 0 | 0
  No symptom, Week 26 | 1 | NA — There is no data because of discontinuation | 1
  Improved, Week 26 | 0 | NA — There is no data because of discontinuation | 0
  Unchanged, Week 26 | 0 | NA — There is no data because of discontinuation | 0
  Worsened, Week 26 | 0 | NA — There is no data because of discontinuation | 0
  No symptom, Week 30 | 1 | NA — There is no data because of discontinuation | 1
  Improved, Week 30 | 0 | NA — There is no data because of discontinuation | 0
  Unchanged, Week 30 | 0 | NA — There is no data because of discontinuation | 0
  Worsened, Week 30 | 0 | NA — There is no data because of discontinuation | 0
  No symptom, Week 34 | 1 | NA — There is no data because of discontinuation | 1
  Improved, Week 34 | 0 | NA — There is no data because of discontinuation | 0
  Unchanged, Week 34 | 0 | NA — There is no data because of discontinuation | 0
  Worsened, Week 34 | 0 | NA — There is no data because of discontinuation | 0
  No symptom, Week 38 | 1 | NA — There is no data because of discontinuation | 1
  Improved, Week 38 | 0 | NA — There is no data because of discontinuation | 0
  Unchanged, Week 38 | 0 | NA — There is no data because of discontinuation | 0
  Worsened, Week 38 | 0 | NA — There is no data because of discontinuation | 0
  No symptom, Week 42 | 1 | NA — There is no data because of discontinuation | 1
  Improved, Week 42 | 0 | NA — There is no data because of discontinuation | 0
  Unchanged, Week 42 | 0 | NA — There is no data because of discontinuation | 0
  Worsened, Week 42 | 0 | NA — There is no data because of discontinuation | 0
  No symptom, Week 46 | 1 | NA — There is no data because of discontinuation | 1
  Improved, Week 46 | 0 | NA — There is no data because of discontinuation | 0
  Unchanged, Week 46 | 0 | NA — There is no data because of discontinuation | 0
  Worsened, Week 46 | 0 | NA — There is no data because of discontinuation | 0
  No symptom, Week 50 | 1 | NA — There is no data because of discontinuation | 1
  Improved, Week 50 | 0 | NA — There is no data because of discontinuation | 0
  Unchanged, Week 50 | 0 | NA — There is no data because of discontinuation | 0
  Worsened, Week 50 | 0 | NA — There is no data because of discontinuation | 0
  No symptom, Week 54 | 1 | NA — There is no data because of discontinuation | 1
  Improved, Week 54 | 0 | NA — There is no data because of discontinuation | 0
  Unchanged, Week 54 | 0 | NA — There is no data because of discontinuation | 0
  Worsened, Week 54 | 0 | NA — There is no data because of discontinuation | 0
  No symptom, at discontinuations | NA — There is no data because of completion | 1 | NA — There is no data because of completion
  Improved, at discontinuations | NA — There is no data because of completion | 0 | NA — There is no data because of completion
  Unchanged, at discontinuations | NA — There is no data because of completion | 0 | NA — There is no data because of completion
  Worsened, at discontinuations | NA — There is no data because of completion | 0 | NA — There is no data because of completion

15. Secondary Outcome: Change From Baseline in Clinical Symptoms Associated With Vascular BD Patients
Description: The investigator assessed the clinical symptoms associated with vascular-BD at each time point of the evaluation in compared to Week 0, in accordance with the categories as "No symptom, Improved, Unchanged or Worsened".
Time Frame: Week 2, 6, 10, then every 4 weeks after Week 14 to Week 54
Measure: Number; unit: participants
Arm/Group | Vascular-BD
Number analyzed (Participants) | 4
participants
  No symptom, Week 2 | 1
  Improved, Week 2 | 2
  Unchanged, Week 2 | 1
  Worsened, Week 2 | 0
  No symptom, Week 6 | 1
  Improved, Week 6 | 2
  Unchanged, Week 6 | 1
  Worsened, Week 6 | 0
  No symptom, Week 10 | 1
  Improved, Week 10 | 2
  Unchanged, Week 10 | 1
  Worsened, Week 10 | 0
  No symptom, Week 14 | 1
  Improved, Week 14 | 2
  Unchanged, Week 14 | 1
  Worsened, Week 14 | 0
  No symptom, Week 18 | 0
  Improved, Week 18 | 4
  Unchanged, Week 18 | 0
  Worsened, Week 18 | 0
  No symptom, Week 22 | 0
  Improved, Week 22 | 3
  Unchanged, Week 22 | 1
  Worsened, Week 22 | 0
  No symptom, Week 26 | 0
  Improved, Week 26 | 3
  Unchanged, Week 26 | 1
  Worsened, Week 26 | 0
  No symptom, Week 30 | 0
  Improved, Week 30 | 4
  Unchanged, Week 30 | 0
  Worsened, Week 30 | 0
  No symptom, Week 34 | 0
  Improved, Week 34 | 3
  Unchanged, Week 34 | 1
  Worsened, Week 34 | 0
  No symptom, Week 38 | 0
  Improved, Week 38 | 4
  Unchanged, Week 38 | 0
  Worsened, Week 38 | 0
  No symptom, Week 42 | 0
  Improved, Week 42 | 4
  Unchanged, Week 42 | 0
  Worsened, Week 42 | 0
  No symptom, Week 46 | 0
  Improved, Week 46 | 4
  Unchanged, Week 46 | 0
  Worsened, Week 46 | 0
  No symptom, Week 50 | 0
  Improved, Week 50 | 4
  Unchanged, Week 50 | 0
  Worsened, Week 50 | 0
  No symptom, Week 54 | 0
  Improved, Week 54 | 4
  Unchanged, Week 54 | 0
  Worsened, Week 54 | 0
  No symptom, Final | 0
  Improved, Final | 4
  Unchanged, Final | 0
  Worsened, Final | 0

ADVERSE EVENTS:
Arm/Group | TA-650
Serious Adverse Events (participants affected / at risk) | 2/18
Other Adverse Events (participants affected / at risk) | 17/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TA-650 (N=18)
Cataract (Eye disorders) | 1
Behcet's syndrome (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TA-650 (N=18)
Bronchitis (Infections and infestations) | 1
Enteritis infectious (Infections and infestations) | 2
Gastroenteritis (Infections and infestations) | 2
Gastroenteritis norovirus (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 4
Periodontitis (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 1
Pulpitis dental (Infections and infestations) | 1
Tinea pedis (Infections and infestations) | 1
Tonsillitis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 5
Depressive symptom (Psychiatric disorders) | 1
Somatoform disorder (Psychiatric disorders) | 1
Dizziness (Nervous system disorders) | 1
Dysaesthesia (Nervous system disorders) | 1
Headache (Nervous system disorders) | 2
Hypoaesthesia (Nervous system disorders) | 1
Intracranial hypotension (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 1
Tension headache (Nervous system disorders) | 1
Conjunctival haemorrhage (Eye disorders) | 1
Dry eye (Eye disorders) | 1
Palpitations (Cardiac disorders) | 1
Behcet's syndrome (Vascular disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Proctalgia (Gastrointestinal disorders) | 2
Cholelithiasis (Hepatobiliary disorders) | 1
Liver disorder (Hepatobiliary disorders) | 1
Acne (Skin and subcutaneous tissue disorders) | 2
Asteatosis (Skin and subcutaneous tissue disorders) | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 1
Dyshidrotic eczema (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2
Muscle rigidity (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1
Malaise (General disorders) | 1
Puncture site reaction (General disorders) | 1
Pyrexia (General disorders) | 2
Antinuclear antibody increased (Investigations) | 2
Double stranded DNA antibody positive (Investigations) | 8
White blood cell count decreased (Investigations) | 1
Administration related reaction (Injury, poisoning and procedural complications) | 1
Arthropod sting (Injury, poisoning and procedural complications) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Excoriation (Injury, poisoning and procedural complications) | 1
Ligament sprain (Injury, poisoning and procedural complications) | 2
Limb injury (Injury, poisoning and procedural complications) | 1
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 1
Tongue injury (Injury, poisoning and procedural complications) | 1
Wound (Injury, poisoning and procedural complications) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other